CLINICAL TRIAL: NCT06365801
Title: Investigation of Acupoint in Irritable Bowel Syndrome Based on Biological Characteristics: A Prospective Cohort Study
Brief Title: Investigation of Acupoint in Irritable Bowel Syndrome Based on Biological Characteristics
Status: Not yet recruiting | Type: Observational
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Xiaomei Shao, Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Other Study IDs: 2022YFC3500401-IBS
Record Dates: First submitted 2024-03-28; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; acupoint; biological characteristics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples and blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers group: There are 50 healthy volunteers in the group.
- IBS group: There are 50 patients in the IBS group.

SUMMARY:
Irritable bowel syndrome (IBS) is a common functional disorder of the digestive system characterized by recurrent abdominal pain associated with bowel movements or changes in bowel habits. Although there are reviews and guidelines for treating IBS, the complexity and diversity of IBS manifestations make treatment difficult. By detecting and exploring the biological characteristics presented by the relevant meridian point reaction, this project clarified the specificity and regularity of the connection between the acupoint and the Zangfu reflected by this phenomenon, and conducted correlation analysis based on the intestinal flora, tryptophan metabolite levels and related scales of patients with IBS.

DETAILED DESCRIPTION:
This study intends to include 50 healthy volunteers and 50 patients with IBS. The study objects are healthy volunteers and patients diagnosed with IBS from the Third Affiliated Hospital of Zhejiang Chinese Medicine University and social recruitment. This study is observational and does not involve randomized methods. At the same time, there is no blindness for subjects, indicators detection and input. The observation indexes were pain sensitivity, thermal radiation characteristics, microcirculation characteristics, biological ultra-weak luminescence, electrical characteristics, intestinal flora characteristics, tryptophan metabolites level and related scales at common acupoints of irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for healthy volunteers:

  1. 18 years old ≤ age ≤75 years old, gender is not limited;
  2. No inflammatory bowel disease, lactose intolerance, intestinal bacterial overgrowth, parasitic infection, drug induced enteritis and other intestinal diseases;
  3. No abdominal pain, frequency of defecation and changes in fecal characteristics in 1 week;
  4. Provide healthy subjects with no obvious abnormalities reported by colonoscopy in the past 1 year;
  5. Healthy subjects who can provide medical examination reports within the past 1 year and have routine physical examination conducted by researchers to confirm that there are no heart and lung diseases, digestive, urinary, blood, endocrine, nervous system and other serious underlying diseases;
  6. No antidiarrheal drugs, antibiotics, gastrointestinal motility drugs or other related drugs affecting clinical studies within 4 weeks;
  7. Clear consciousness, can complete normal communication;
  8. Understands and is willing to comply with the research protocol and sign the informed consent.
* Inclusion criteria for IBS patients:

  1. Patients who can provide colonoscopy report in the past 1 year and meet the Rome IV standard of irritable bowel syndrome and TCM syndrome differentiation type;
  2. Provide medical examination reports within the past 1 year to confirm patients without digestive, circulatory, respiratory, urinary, reproductive, endocrine, nervous system and other malignant tumors and serious underlying diseases;
  3. 18 years old ≤ age ≤75 years old, gender is not limited;
  4. No antidiarrheal drugs, antibiotics, gastrointestinal motility drugs or other related drugs that affect clinical studies have been taken within 4 weeks;
  5. Clear consciousness, can complete normal communication;
  6. Understands and is willing to comply with the research protocol and sign the informed consent.

Exclusion Criteria:

* Exclusion criteria for healthy volunteers:

  1. Those who have mental illness, alcohol dependence or a history of drug abuse and cognitive impairment are unable to cooperate with the examination and understanding of the subject;
  2. Female volunteers who are pregnant or lactating, or in ovulation and menstruation period;
  3. Volunteers with current abnormal body temperature;
  4. Subjects currently participating in other clinical trials.
* Exclusion criteria for patients with IBS:

  1. Those who have mental illness, alcohol dependence or a history of drug abuse and cognitive impairment are unable to cooperate with the examination and understanding of the subject;
  2. Pregnant or lactating women or female subjects in ovulation and menstruation period;
  3. Patients with inflammatory bowel disease, lactose intolerance, intestinal bacterial overgrowth, parasitic infections, drug-induced enteritis and other intestinal diseases;
  4. Patients with intestinal diseases such as functional constipation, functional diarrhea, opioid-induced constipation, and non-specific functional bowel disease;
  5. Patients with functional gastrointestinal diseases such as functional dyspepsia, functional heartburn, central abdominal pain syndrome;
  6. Patients with current abnormal body temperature;
  7. Participants who are currently participating in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study targets IBS patients and healthy volunteers, among whom IBS patients are required to meet the Rome IV standard for IBS and the Expert Consensus on the Diagnosis and Treatment of IBS in Chinese Medicine (2017).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain sensitivity | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  Select the measurement point, place the probe of the handheld pain threshold testing instrument vertically on the pain measurement point, slowly and steadily press, and stop the pressure when the subject feels pain (or the subject can stop the pressure). At this point, the reading on the monitor is the subject's pain threshold. After the measurement is completed, press the zero button to measure the next point or the next subject.
Thermal radiation characteristics | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  The NEC R550 infrared thermal imager and the InfRec Analyzer NS9500 computer software were used to store and save the infrared thermal images taken, and the temperature data were analyzed, the temperature values of relevant acupoints in corresponding coordinates were extracted, and the average temperature values of acupoints in the 6 infrared thermal images were calculated as their basic temperatures.
Microcirculation characteristics | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  The PeriCam PSI laser speckle imager was adopted to store and record the speckle imaging images and curves with the support of PIM Soft computer software, and the blood flow data was analyzed, the blood flow values of the corresponding acupoints were extracted, and the average perfusion volume of the acupoints within 2 minutes was calculated as the perfusion volume index.
Electrical characteristics | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  Meridian point resistance meter was used to measure the point resistance, each point was detected for 5 minutes, the data was stored and analyzed by excel2019, the relative resistance value of the corresponding point was extracted, and the average resistance value of the point was calculated within 5 minutes.
Biological ultra-weak luminescence | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  It is divided into the UPE detection system of photomultiplier tube (PMT) and the UPE image acquisition system of charge coupled device (CCD).PMT: The data of each measurement point is the self-luminous intensity of the subject per second.CCD: The image acquisition software Andor Solis is used to store the captured CCD image, analyze the ultra-weak luminescence data of the acquisition site, and extract the average value of the ultra-weak luminescence of the corresponding position as its basic value.

SECONDARY OUTCOMES:
Intestinal flora | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  the distribution structure and biodiversity of intestinal flora
Tryptophan metabolites | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  the levels of L-tryptophan and 5-hydroxytryptophan (5-HT), 5-hydroxyindoleacetic acid (5-HIAA), Kyine (KYN), Kyine acid (KYNA), quinolinic acid (QA) and other related metabolites in plasma
Bristol Fecal Traits Grading Scale | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  Based on patient reports of at least 14 days, the "25% rule" was used (that is, fecal traits were recorded according to the major abnormal bowel habits in the presence of abnormal bowel movements, combined with the Bristol classification table to determine which subtype they belonged to).
Severity of IBS (IBS-SSS) | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  The scale includes 5 aspects, including the degree of abdominal pain, the frequency of abdominal pain, the degree of abdominal distension, the satisfaction of defecation and the impact on life. The full score of each item is 100 points, and the total score is 500 points. Evaluation criteria: 1) Normal :≤75 points; 2) Mild :76 ~ 175 points; 3) Moderate :176 ~ 300 points; 4) Heavy: > 300 points.
IBS Quality of Life (IBS-QOL ) | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  The scale contained 34 items in 8 dimensions including restlessness, activity restriction, body image, health concern, dietary restriction, social and sexual disturbance, and interpersonal relationship. Patients were given descriptive statements of the past 1 month (30 days) recall period, and were evaluated using five rating options of "none, mild, moderate, severe, and very severe." "None" is rated 1 point, "mild" 2 points, "moderate" 3 points, "severe" 4 points, and "very severe" 5 points. All items are given a total score to calculate the total, with higher scores indicating better health-related quality of life.
TCM Constitution Survey | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  The physical fitness scale refers to the Traditional Chinese Medicine Physical Fitness Survey Scale compiled by Professor Wang Qi, which is widely used in clinical practice at present. It includes nine types of physical fitness, of which only peace and quality are normal physical fitness, and the rest are biased physical fitness. The physical fitness calculation method is as follows: Firstly, the original score of each physical fitness subscale is calculated (that is, the score of each item of each subscale is added together), and then the physical fitness conversion score is calculated according to the original score. Conversion score = (original score - number of entries)/(number of entries *4) * 100.
Gastrointestinal Symptoms Rating Scale (GSRS) | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  Gastrointestinal Symptom Rating Scale (GSRS) consists of 15 self-rated items, including gastrointestinal symptom intensity, seizure frequency, seizure duration and impact on daily life, with a score of 1-7 for each item. A higher total score indicates more severe gastrointestinal symptoms.
Self-Rating Anxiety Scale (SAS) | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  SAS contains 20 items reflecting the subjective feeling of anxiety, and each item is graded according to the frequency of symptoms, of which 15 are positive scores and 5 are reverse scores. (5, 9, 13, 17, and 19 are inverted scores.) According to the results of the Chinese norm, the cut-off value of SAS standard score is 50 points, in which 50 ~ 59 is classified as mild anxiety, 60 ~ 69 is classified as moderate anxiety, and more than 69 is severe anxiety.
Self-Rating Depression Scale (SDS) | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  SDS contains 20 items reflecting the subjective feeling of depression, and each item is divided into four grades according to the frequency of symptoms, of which 10 are positive scores and 10 are reverse scores. According to the results of Chinese norm, the cut-off value of SDS standard score was 53 points, of which 53 ~ 62 were classified as mild depression, 63 ~ 72 was classified as moderate depression, and 72 or more were classified as severe depression.
Pittsburgh Sleep Quality Index (PSQI) | the baseline and 4 times during the follow-up period (1st month, 2nd month, 4th month and 6th month after enrollment)
  PSQI was used to assess the sleep quality of the participants in the last 1 month. It consists of 19 reviews and 5 other reviews, of which the 19th review and 5 other reviews do not participate in the scoring, only 18 reviews that participate in the scoring are introduced here. The 18 items were composed of 7 components, each component was scored according to 0~ 3 levels, and the cumulative score of each component was the PSQI total score, the total score range was 0~2l, the higher the score, the worse the sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University

IPD SHARING:
Plan to Share IPD: No